CLINICAL TRIAL: NCT07286695
Title: A Multicenter, Open-label, Randomized Controlled Study of Fruquintinib Combined With Trifluridine/Tipiracil Versus Bevacizumab Combined With Trifluridine/Tipiracil in the Treatment of Patients With Advanced Metastatic Colorectal Cancer Who Failed Standard Chemotherapy
Brief Title: Fruquintinib Combined With Trifluridine/Tipiracil Versus Bevacizumab Combined With Trifluridine/Tipiracil for Advanced Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, AIPING ZHOU, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C138
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Cancer (CRC); Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine; tipiracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fruquintinib and trifluridine/tipiracil (Experimental)
  Interventions: Drug: Fruquintinib Combined With trifluridine/tipiracil
- Bevacizumab and trifluridine/tipiracil (Active Comparator)
  Interventions: Drug: Bevacizumab combined with trifluridine/tipiracil

INTERVENTIONS:
Drug: Fruquintinib Combined With trifluridine/tipiracil — Experimental arm: Fruquintinib: 4mg once daily for 21 days on/7 days off, every 28 days; Trifluridine/tipiracil: taken at a recommended dose (based on the results of the safety run-in phase) each time orally twice a day on days 1-5 and 8-12, every 28 days.
  Arms: Fruquintinib and trifluridine/tipiracil
Drug: Bevacizumab combined with trifluridine/tipiracil — Active Comparator: Bevacizumab: 5 mg /kg, intravenously on days 1,15, every 28 days; Trifluridine/tipiracil: 35 mg/m²orally twice a day on days 1-5 and 8-12, every 28 days.
  Arms: Bevacizumab and trifluridine/tipiracil

SUMMARY:
Fruquintinib, as a standard treatment for refractory metastatic colorectal cancer (mCRC), has attracted increasing research efforts to explore its innovative strategies in combination with chemotherapy. Trifluridine/tipiracil plus bevacizumab is also a standard treatment for mCRC. This study aims to explore the efficacy and safety of fruquintinib combined with trifluridine/tipiracil versus bevacizumab combined with trifluridine/tipiracil in the treatment of patients with advanced metastatic colorectal cancer who failed standard chemotherapy.

DETAILED DESCRIPTION:
Phase II study comprises a safety run-in stage, and a randomized treatment stage.

Phase II (safety run-in stage): It aims to evaluate the safety and tolerability of combination therapy-comprising trifluridine/tipiracil and fruquintinib. Trifluridine/tipiracil was administered at a descending dose level starting from 35 mg/m² each time alongside fixed dose of fruquintinib in mCRC patients who have previously received first-line oxaliplatin and irinotecan-based therapy, or have failed at least two lines of standard chemotherapy regimens.

Phase II (randomized treatment stage): Upon determination of the recommend dose of trifluridine/tipiracil based on prior data, a randomized controlled study will be conducted in mCRC patients who have previously received first-line oxaliplatin and irinotecan-based therapy, or have failed at least two lines of standard chemotherapy regimens. Patients will be randomly assigned to two arms: experimental arm: Fruquintinib and trifluridine/tipiracil; active comparator arm: Bevacizumab and trifluridine/tipiracil.

ELIGIBILITY:
Inclusion Criteria:

* Have a full understanding of this study and voluntarily sign the informed consent form;
* Aged 18-75 years old (including 18 and 75 years old);
* Diagnosed with advanced metastatic colorectal adenocarcinoma by histopathological examination;
* Patients who have previously received first-line oxaliplatin and irinotecan treatment, or have received and failed at least two lines of standard chemotherapy regimens. These standard treatment regimens must include fluoropyrimidine-based drugs, oxaliplatin and irinotecan (with or without bevacizumab or cetuximab). Treatment failure is defined as disease progression occurring during treatment or within 3 months after the last treatment, or intolerable toxic side effects. Each line of treatment must include one or more chemotherapy drugs administered for ≥1 cycle; if recurrence or metastasis occurs during adjuvant/neoadjuvant treatment or within 6 months after completion of adjuvant/neoadjuvant treatment, the adjuvant/neoadjuvant treatment is considered a failure of first-line chemotherapy for advanced disease;
* Have previously received bevacizumab treatment;
* Must have at least one clear measurable lesion that meets the requirements of the Response Evaluation Criteria in Solid Tumors (RECIST 1.1);
* ECOG performance status of 0-1;
* Expected survival time ≥12 weeks;
* Within 7 days before enrollment, the function of important organs must meet the following requirements (the use of any blood components and cell growth factors within 14 days before enrollment is not allowed):

Absolute neutrophil count ≥1.5×10⁹/L; Platelets ≥80×10⁹/L; Hemoglobin ≥8g/dL; Total bilirubin ≤1.5×ULN (upper limit of normal); ALT (alanine aminotransferase) and AST (aspartate aminotransferase) ≤2.5×ULN (for patients with liver metastasis, ≤5×ULN); Serum creatinine ≤1.5×ULN, and estimated glomerular filtration rate ≥50ml/min; International Normalized Ratio (INR) ≤1.5 or activated partial thromboplastin time (APTT) ≤1.5×ULN;

• Good compliance and willingness to cooperate with follow-up.

Exclusion Criteria:

* Unable to comply with the study protocol or procedures;
* Previous treatment with TAS-102 or vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitors (TKIs) (e.g., anlotinib, apatinib, etc.);
* Participation in other drug clinical trials within 4 weeks before enrollment;
* Have received or is currently receiving other systemic anti-tumor treatments within 4 weeks prior to enrollment;
* Patients with currently uncontrolled hypertension (defined as systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg) despite medication;
* Patients with current diseases or conditions that affect drug absorption, or patients unable to take oral medications;
* Patients with active gastrointestinal diseases such as active gastric and duodenal ulcers, ulcerative colitis, active bleeding from unresected tumors, or other conditions judged by the investigator to potentially cause gastrointestinal bleeding or perforation;
* History of arterial thrombosis or deep vein thrombosis within 6 months before enrollment;
* Patients with evidence or medical history of significant bleeding tendency within 2 months before enrollment, such as melena, hematemesis, hemoptysis, fecal occult blood test (FOBT) result of ++ or above (for patients with FOBT result of + and existing primary lesions, gastroscopy must be performed to rule out bleeding or ulcers before enrollment);
* History of stroke and/or transient ischemic attack within 12 months before enrollment; presence of cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months before enrollment; congestive heart failure of New York Heart Association (NYHA) class >2; ventricular arrhythmias requiring medication; left ventricular ejection fraction (LVEF) <50% (confirmed by echocardiography);
* History of other malignant tumors within the past 5 years, except for fully treated basal cell carcinoma or squamous cell carcinoma of the skin, carcinoma in situ of organs such as the cervix, early non-invasive lung cancer, and non-muscle-invasive bladder cancer;
* Clinically uncontrolled active infections, such as acute pneumonia, active hepatitis B or C (for patients with a history of hepatitis B virus infection, regardless of medication control, hepatitis B virus DNA ≥1×10⁴ copies/mL or >2000 IU/mL);
* Pregnant women (positive pregnancy test before medication administration) or lactating women;
* Urinalysis showing urine protein ≥2+, or 24-hour urine protein quantitation >1.0g;
* Patients deemed unsuitable for enrollment in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | About 3 years
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | About 3 years
  ORR was defined as the percentage of patients with a best overall response of complete response (CR) or partial response (PR) per RECISTv1.1.
Disease control rate (DCR) | About 3 years
  DCR was defined as the percentage of patients with a best overall response of confirmed complete or partial response, or stable disease (CR+ PR + SD) per RECISTv1.1.
Overall survival (OS) | About 3 years
  OS was defined as the time from the date of randomization to the date of death due to any cause.
Adverse Events (AE) | About 3 years
  Adverse Events (AE) as assessed by CTCAE v5.0, including serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD shared with other researchers will include the study protocol.
Supporting Information: Study Protocol
Time Frame: IPD will be made available 12 months after the primary publication of the study's main results.
Access Criteria: Eligible recipients must submit an approved research proposal and sign a data use agreement.

REFERENCES:
- [Result] Nukatsuka M, Fujioka A, Nagase H, Tanaka G, Hayashi H. Evaluation of a Novel Combination Therapy, Based on Trifluridine/Tipiracil and Fruquintinib, against Colorectal Cancer. Chemotherapy. 2023;68(2):102-110. doi: 10.1159/000528867. Epub 2023 Jan 9. PMID 36623495
- [Result] Zou J, Wang Y, Xu J, Li J, Wang T, Zhang Y, Bai Y. A Retrospective Study of Trifluridine/Tipiracil with Fruquintinib in Patients with Chemorefractory Metastatic Colorectal Cancer. J Clin Med. 2023 Dec 21;13(1):57. doi: 10.3390/jcm13010057. PMID 38202064